CLINICAL TRIAL: NCT01737333
Title: A Multicenter, Multinational, Randomized Study of Standard vs. Patient-Adapted Protocols in Multidetector Computed Tomography (MDCT) of the Chest, Abdomen, Liver or Aorta
Brief Title: Multidetector Computed Tomography (MDCT) Tailored Protocol
Status: Completed | Type: Observational
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: IOPM-101
Record Dates: First submitted 2012-11-20; First posted 2012-11-29 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Patients Undergoing Contrast Enhanced Multidetector Computed Tomography of the Chest, Abdomen, Liver or Aorta for Any Diagnostic Cause

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Collection of data from different sites regardless of whether they use standard or tailored protocols for the application of high concentration iodinated contrast agents to assess if the individually patient-adapted protocols result in a similar diagnostic image quality.

DETAILED DESCRIPTION:
To record technical information and compare image quality regarding routine MDCT procedures with contrast administration using a tailored contrast injection and radiation dose protocol. The hypotheses are that the tailored protocols lead to a lower applied mean radiation dose compared to the use of standard protocols and will provide a more standardized contrast dose per patient size without impairing diagnostic quality.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Scheduled to undergo contrast enhanced MDCT of the abdomen, liver, aorta, or chest
* Provides written informed consent

Exclusion Criteria:

* Previously enrolled and completed the study
* Known allergy to iodinated contrast media
* Pregnancy or lactation
* Clinically unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing MDCT of the abdomen, liver, chest or aorta and receiving high iodinated contrast agents
Sampling Method: Probability Sample
Enrollment: 1493 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic Quality | Immediately after the single injection of contrast agent
  Images are to be assessed according to the following scale: 0=Uninterpretable (Image quality severely affected by motion artifacts or technical reasons; need to repeat the examination); 1=Insufficient (Impaired image quality precludes adequate diagnostic assessment because of severe image noise or insufficient contrast enhancement; need to repeat the examination); 2=Adequate (Image quality in terms of noise and contrast enhancement does not interfere with sufficient diagnostic assessment; delineation of small structures may be suboptimal); or 3=Good (Absent or minimal image noise and good contrast enhancement allow adequate diagnostic assessment with clear delineation of even small structures).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Krix, M.D., Study Director — Bracco Diagnostics, Inc
Locations (2):
- Department of Radiology Carolinas Medical Center, Charlotte, North Carolina, United States
- Oepedale Niguarda, Milan, Italy